CLINICAL TRIAL: NCT02833961
Title: DIFFUSION SPECTROSCOPY AND IMAGING IN ACUTE STROKE
Brief Title: Diffusion Spectroscopy in Stroke
Acronym: ISIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: C16-04; 2016-A00362-49 (Registry Identifier: IDRCB)
Record Dates: First submitted 2016-06-15; First posted 2016-07-14 (Estimated); Last update posted 2025-09-03 (Actual); Status verified 2021-08

CONDITIONS: ISCHEMIC STROKE
MeSH Terms: conditions — Ischemic Stroke | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- ISCHEMIC STROKE (Experimental): ischemic stroke admitted in the Pitié Salpêtrière Stroke unit in Paris
  Interventions: Device: Magnetic resonance imaging
- HEALTHY SUBJECTS (Active Comparator): Age and gender-matched healthy volunteers
  Interventions: Device: Magnetic resonance imaging

INTERVENTIONS:
Device: Magnetic resonance imaging

SUMMARY:
Cerebral vascular disorder is one of the most fatal diseases despite current advances in medical science. The large number of negative clinical trials on neuroprotection in acute stroke is a pointer to the fact that translating better understanding of the pathogenesis and pathophysiology to clearly beneficial treatment strategies remains a daunting task. This project aims at elucidating the plausible biophysical events that affect water and metabolite diffusion in brain tissue after ischemia, by combining the information provided by two advanced methods of magnetic resonance (MR) diffusion imaging: diffusional kurtosis imaging and diffusion-weighted spectroscopy.

Diffusion weighted imaging (DWI) has been established as a major tool for the early detection of stroke. However, information obtained using conventional DWI may be incomplete. Diffusional kurtosis (K) is a quantitative measure of the complexity or heterogeneity of the microenvironment in white and grey matter, which offers complementary information and may potentially be a more sensitive biomarker for probing pathophysiological changes. In addition, to gain more specific insights into molecular mobility in the intracellular environment, it is beneficial to assess the diffusion properties of metabolites, such as N-acetylaspartate (NAA), creatine and phosphocreatine (Cr), and choline containing compounds (Cho). Assessment of metabolite diffusion changes by diffusion-weighted spectroscopy (DWS) provides information specific to the intracellular environment. In particular, thanks to the specific compartmentation of NAA almost exclusively in neurons and of Cho in glial cells, the diffusion properties of these metabolites may provide specific insights into the pathological processes occurring independently in the two cell types. In addition, measuring a temporal profile of diffusion coefficient of these compounds may help clarify underlying pathophysiological changes in neuronal cells during acute ischemia.

With the help of these two advanced methods, a proof-of-concept trial is proposed on 24 healthy subjects and 24 ischemic stroke patients. Ischemic stroke patients will be scanned three times with a 3T MR scanner (before day 10 post-stroke, around week 4 and 3 months), in order to extract diffusion kurtosis imaging (DKI) and DWS metrics and understand the dynamics of the cellular mechanisms at play in cerebral ischemia. The goal of this study is to investigate neuronal and glial metabolite diffusion changes at different time points after ischemic stroke, in both infarcted and non-infarcted hemispheres. The aim is to get non-invasively important information on the evolution of the cellular damage in this disease, and possibly distinguishing between neuronal and glial processes (by measuring the metrics extracted for these two sequences), as well as on the different mechanisms leading to metabolite diffusion changes in the two brain areas, thus providing a great impact on the strategy of treatment for patients with cerebral infarction.

ELIGIBILITY:
Inclusion Criteria:

first-ever infarct lesion Infarct volume > 8 cm3 written consent French social security

Exclusion Criteria:

age <18 or >80 years contraindication to MRI Life-threatening disease that could compromise the follow-up Pregnant and breast-feeding women Patients under a legal gardian

We will also include 24 healthy subjects for comparison with no history of neurological disease.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-07-28 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
ADC measurements (in mm2/second) of metabolites within the ischemic lesion | up to 14 days

SECONDARY OUTCOMES:
Relative change of the ADC values (in %) of the metabolites over time | 1 and 3 months
Diffusivity measure within the ischemic lesion (in mm2/second). | up to14 days
Relative change of the diffusivity measure values (in %) of water over time | 1 and 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institut du cerveau et de la moelle, Hôpital Pitié-Salpétrière, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ashktorab K, Janecke JW, Becchetti FD. Beta decay of 187Re and cosmochronology. Phys Rev C Nucl Phys. 1993 Jun;47(6):2954-2960. doi: 10.1103/physrevc.47.2954. No abstract available. PMID 9968771
- [Derived] Genovese G, Diaz-Fernandez B, Lejeune FX, Ronen I, Marjanska M, Yahia-Cherif L, Lehericy S, Branzoli F, Rosso C. Longitudinal Monitoring of Microstructural Alterations in Cerebral Ischemia with in Vivo Diffusion-weighted MR Spectroscopy. Radiology. 2023 Mar;306(3):e220430. doi: 10.1148/radiol.220430. Epub 2022 Nov 1. PMID 36318030